CLINICAL TRIAL: NCT00676676
Title: Effects of Testosterone in Women With Depression: A Pilot Study
Brief Title: Effects of Testosterone in Women With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007p000348
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Testosterone (Active Comparator): Testosterone patch delivering 300mcg daily for 8-weeks.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone atch delivering 300mcg daily for 8-weeks

SUMMARY:
The purpose of the study is to determine whether adding a low dose of testosterone to current antidepressant therapy improves depression and fatigue in women who remain depressed despite necessary adequate doses of anti-depressants. Testosterone will be given over an 8-week period.

Testosterone is a hormone that occurs naturally in the body. In women it comes from the ovaries and adrenal glands and is found in amounts that are ten to twenty times lower than in men.

In early research studies, testosterone has been shown to have some antidepressant effects in the following groups of subjects:

* Women with anorexia nervosa
* Women who have low testosterone levels because their pituitary glands do not work
* Men with Selective Serotonin Reuptake Inhibitor (SSRI)-resistant depression.

However, testosterone administration in women with SSRI or Serotonin-norepinephrine reuptake inhibitor (SNRI) -resistant depression has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-75
* Written informed consent
* Meet Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria (by Structured Clinical Interview for DSM-IV (SCID)) for Major Depressive Disorder
* Meet DSM-IV criteria for a current major depressive episode, as assessed by SCID
* Montgomery-Asberg Depression Rating Scale (MADRS) greater than or equal to 16 at baseline visit
* Currently treated with SSRI or SNRI, with or without adjunctive therapy, at an adequate dose (see adequate dose table below) for at least six weeks

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
* Serious suicide or homicide risk, as assessed by evaluating clinician
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic (including uncontrolled seizure disorder)
* Substance use disorder active within last six months
* Psychotic features (current episode or lifetime), as assessed by SCID
* Laboratory evidence of untreated hypothyroidism
* If treated hypothyroidism, significant change in levo-thyroxine dose within the prior three months
* If receiving oral estrogen therapy, including oral contraceptives or transdermal estrogen therapy, significant change in dose in the prior three months
* Use of androgens or androgen precursors, including testosterone, Dehydroepiandrosterone (DHEA) and methyltestosterone, within the prior three months
* Any investigational psychotropic drug within the last two weeks
* In the judgment of the study clinician, unlikely to be able to participate safely throughout the study period (three or more episodes of self-harm in the past year, documented history of poor treatment adherence, or frequent missed appointments (greater than 50%) in the past year)
* Alanine aminotransferase (ALT) greater than 1.5 times the upper limit of normal.
* Creatinine greater than 1.5 times upper limit of normal
* History of a hormone-responsive cancer
* History of congestive heart failure
* MADRS greater than 31

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachsuetts General Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone: Testosterone Patch 300mcg replaced every 3-4 days
Period: Overall Study
Arm/Group | Testosterone
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Scale
Description: the MADRS is a diagnostic questionnaire that is used to measure the severity of depressive episodes in patients with mood disorders. The minimum and maximum values are 0 and 60 respectively (higher scores are more severe).
Time Frame: Baseline, 2-week, 8-week
Population: This was a pilot protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone
Number analyzed (Participants) | 9
units on a scale
  Baseline visit | 25.9 (4.6)
  2-week visit | 14.7 (8.4)
  8-week visit | 15.2 (10.9)
Statistical Analysis 1: Comparison: Testosterone; Baseline versus 2-week; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Testosterone; Baseline versus 8-week; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8-weeks
Arm/Group | Testosterone
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=9)
erythema at testosterone patch site (Skin and subcutaneous tissue disorders) | 1 (1)
oily skin/acne (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes